CLINICAL TRIAL: NCT06236529
Title: Supporting Patient Activation for Self-Management of Chronic Low Back Pain With a Targeted Intervention Based on Key Influencing Characteristics
Brief Title: Self-Management of Chronic Low Back Pain: Targeting Patient Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00313911
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Chronic Low-back Pain; Patient Activation
Keywords: Self-management; Nurse-led; Web-based
MeSH Terms: conditions — Patient Participation | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors were masked to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants receive no intervention.
- Self-management program (SMP) (Active Comparator): Participants engage in a nurse-led evidence-based web-enabled group self-management class for 6 weeks.
  Interventions: Behavioral: Self-management program
- Self-management program (SMP) with Health Behavior Change Counseling (HBCC) (Experimental): Participants engage in a nurse-led evidence-based web-enabled group self-management class for 6 weeks and receive three telephone-based health behavioral change counseling sessions based on the principles and practices of motivational interviewing.
  Interventions: Behavioral: Health Behavior Change Counseling; Behavioral: Self-management program

INTERVENTIONS:
Behavioral: Health Behavior Change Counseling — A telephone-based intervention employing principles and practices of motivational interviewing.
  Arms: Self-management program (SMP) with Health Behavior Change Counseling (HBCC)
Behavioral: Self-management program — An evidence-based 6-week SMP led by a registered nurse. The SMP was based on the Arthritis Self-Management Program and the Chronic Disease Self-Management Program.
  Arms: Self-management program (SMP); Self-management program (SMP) with Health Behavior Change Counseling (HBCC)

SUMMARY:
Patients with chronic low back (cLBP) pain report reduced physical function and ability to participate in social roles and are more likely to use opioid pain medications. While self-management interventions have been shown to support these patients, effectiveness has been limited due to poor patient engagement. "Patient activation" encompasses the skills, knowledge, and motivation that a person has to manage the person's health. Supporting patient activation may improve the effectiveness of self-management for cLBP.

In this single-masked pilot study of adults with cLBP, patients were randomized to receive either no intervention (control) or 6 weekly sessions of an evidence-based web-based self-management program (SMP) with or without health behavior change counseling (HBCC) using motivational interviewing. Participants were assessed at baseline and at 12 and 26 weeks using the Patient Activation Measure, Oswestry Disability Index and Patient-Reported Outcomes Measurement Information System (PROMIS) physical function, social role participation, and pain interference. The investigators assessed acceptability and feasibility based on recruitment, session attendance, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years of age)
* Seen in primary or specialty care practice for non-specific low back pain
* Chronic low back pain per the NIH Task Force on Research Standards for cLBP
* Worst back pain of at least 4/10 points
* Oswestry disability index of at least 24%
* English speaking

Exclusion Criteria:

* History of lumbar spine decompression/laminectomy or fusion surgery in the past 6 months
* Possible non-musculoskeletal cause for LBP symptoms diagnosis at baseline
* "Red flag" LBP diagnosis in the previous 6 months (e.g., cauda equina syndrome, osteomyelitis, or spinal neoplasm)
* Neurological disorder resulting in moderate to severe movement dysfunction
* Presence of any psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Acceptability of research | Baseline
  Acceptability - at least 50% of individuals approached agree to eligibility screening for the study, having at least 30% of those who were deemed eligible for the study agree to participate
Feasibility of study | Baseline
  Feasibility - (1) having at least 80% of enrolled participants attend at least 3 of the 6 scheduled self-management program sessions; and (2) having a loss to follow-up rate of < 20% of enrolled participants over the 26-week study

SECONDARY OUTCOMES:
Patient Activation Measure (PAM) score | 12 weeks
  The Patient Activation Measure (PAM) is a 13-item instrument where patients are provided 5 response options, ranging from "strongly agree" to "strongly disagree." Based on their answers, patients were assigned a numerical score ranging from 0 (no activation) to 100 (highest activation), and the score was used to stratify patients into 1 of 4 stages of activation: stage 1 (believes taking an active role is important), stage 2 (has the confidence and knowledge to take action), stage 3 (takes action), and stage 4 (stays the course under stress)
Oswestry Disability Index (ODI) score | 12 weeks
  Pain-related disability was assessed using the ODI, a 10-item measure of low back pain-related disability that evaluates the current effect of a patient's low back pain on various aspects of daily living. ODI scores range from 0 to 100, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Skolasky, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skolasky RL, Nolan S, Pierre R, Vinch P, Taylor JL. Nurse-led web-based self-management program to improve patient activation and health outcomes in patients with chronic low back pain: an acceptability and feasibility pilot study. BMC Nurs. 2024 Jul 31;23(1):524. doi: 10.1186/s12912-024-02155-w. PMID 39085831